CLINICAL TRIAL: NCT05567952
Title: AN INTERVENTIONAL, EFFICACY AND SAFETY, PHASE 2, RANDOMIZED, DOUBLE-BLIND, 2-ARM STUDY TO INVESTIGATE A REPEAT 5-DAY COURSE OF NIRMATRELVIR/RITONAVIR COMPARED TO PLACEBO/RITONAVIR IN PARTICIPANTS AT LEAST 12 YEARS OF AGE WITH REBOUND OF COVID-19 SYMPTOMS AND RAPID ANTIGEN TEST POSITIVITY
Brief Title: A Study to Learn About a Repeat 5-Day Treatment With the Study Medicines (Called Nirmatrelvir/Ritonavir) in People 12 Years Old or Older With Return of COVID-19 Symptoms and SARS-CoV-2 Positivity After Finishing Treatment With Nirmatrelvir/Ritonavir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C4671042; 2022-002827-36 (EudraCT Number)
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Coronavirus disease 2019 (COVID-19); COVID-19 rebound; Paxlovid; Nirmatrelvir
MeSH Terms: conditions — COVID-19; COVID-19 rebound | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- nirmatrelvir plus ritonavir for 5 days (Experimental): Nirmatrelvir (2 tablets) plus ritonavir (1 capsule) will be given by mouth every 12 hours for 5 days
  Interventions: Drug: nirmatrelvir; Drug: ritonavir
- placebo plus ritonavir for 5 days (Other): placebo (2 tablets) plus ritonavir (1 capsule) will be given by mouth every 12 hours for 5 days
  Interventions: Drug: ritonavir; Drug: placebo for nirmatrelvir

INTERVENTIONS:
Drug: nirmatrelvir — Participants will receive 2 tablets of nirmatrelvir every 12 hours
  Arms: nirmatrelvir plus ritonavir for 5 days
Drug: ritonavir — Participants will receive 1 capsule of ritonavir every 12 hours
Drug: placebo for nirmatrelvir — Participants will receive 2 tablets of placebo for nirmatrelvir every 12 hours. A placebo does not have any medicine in it but looks just like the medicine being studied.
  Arms: placebo plus ritonavir for 5 days

SUMMARY:
The purpose of this study is to learn about the safety and effects of nirmatrelvir/ritonavir for the potential treatment of COVID-19 rebound.

The study is seeking participants who:

* Have completed treatment with nirmatrelvir/ritonavir
* Have a rebound in COVID-19 symptoms
* Are SARS-CoV-2 (COVID-19) positive

All study medications will be taken 2 times a day by mouth for 5 days. The first dose of study medication is taken at the study clinic and the rest at home.

We will examine the experiences of people receiving the study medicines to those who do not. This will help us determine if the study medicines are safe and effective.

People taking part will be in this study for about 24 weeks. Enrolled participants will need to visit the study clinic at least 8 times during the study.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of nirmatrelvir/ritonavir treatment with patient-reported 100% compliance. Symptom alleviation or resolution in COVID-19 signs/symptoms followed by a worsening (rebound) of signs/symptoms after completing an initial 5-day course of nirmatrelvir/ritonavir
* Onset of rebound in COVID-19 symptoms within 2 weeks (14 days) after the completion of the initial 5-day course of nirmatrelvir/ritonavir.
* Onset of rebound in signs/symptoms attributable to COVID-19 within 48 hours prior to randomization and ≥1 sign/symptom attributable to COVID-19 present on the day of randomization.
* SARS-CoV-2 infection as determined by rapid antigen testing within 24 hours prior to randomization
* At least 1 characteristic or underlying medical condition associated with an increased risk of developing severe illness from COVID-19.

Exclusion Criteria:

* Current need for hospitalization, hospitalized for the COVID-19 infection or anticipated need for hospitalization within 24 hours after randomization
* History of severe chronic liver disease
* Receiving dialysis or have known age-specific estimated glomerular filtration rate (eGFR) or estimated creatinine clearance (eCrCl) <30 mL/min/1.73 m2 at screening as measured by a serum creatinine point of care device
* Oxygen saturation of <92% on room air obtained at rest within 24 hours prior to randomization
* Immunocompromised.
* Current use of any prohibited concomitant medication(s)
* Females who are pregnant and <14 weeks gestation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (67):
  - The Institute for Liver Health dba Arizona Clinical Trials, Mesa, Arizona
  - Abby's Research institute, Phoenix, Arizona
  - Epic Medical Research - Surprise, Surprise, Arizona
  - Smart Cures Clinical Research, Anaheim, California
  - Hope Clinical Research, Inc., Canoga Park, California
  - Ascada Health PC dba Ascada Research, Fullerton, California
  - Ascada Research, Fullerton, California
  - Paradigm Clinical Research Centers, Inc, La Mesa, California
  - CVS Health - 8876 - Long Beach, Long Beach, California
  - Carbon Health - North Hollywood - NoHo West, North Hollywood, California
  - Paradigm Clinical Research Centers, Inc, Wheat Ridge, Colorado
  - Emerson Clinical Research Institute - Washington - Connecticut Avenue, Washington D.C., District of Columbia
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Palm Harbor Dermatology PA d/b/a TrueBlue Clinical Research, Brandon, Florida
  - Herco Medical and Research Center Inc, Coral Gables, Florida
  - NeoClinical Research, Hialeah, Florida
  - Sweet Hope Research Specialty, Inc, Hialeah, Florida
  - Unlimited Medical Research Group LLC, Hialeah Gardens, Florida
  - Asclepes Research Center - Spring Hill, Lutz, Florida
  - LCC Medical Research Institute, Miami, Florida
  - Premium Medical Research Corp, Miami, Florida
  - Global Health Clinical Trials, Miami, Florida
  - South Florida Research Center, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Innova Pharma Research, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Reed Medical Research, Miami, Florida
  - Kendall South Medical Center, Miami, Florida
  - Pro-Care Research Center, Corp., Miami Gardens, Florida
  - Omega Research Orlando, Orlando, Florida
  - NAPA Research, Pompano Beach, Florida
  - Asclepes Research Center - Spring Hill, Spring Hill, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - Theia Clinical Research - 5th Avenue North, St. Petersburg, Florida
  - Palm Harbor Dermatology PA d/b/a TrueBlue Clinical Research, Tampa, Florida
  - Santos Research Center, Tampa, Florida
  - Clinical Site Partners, LLC dba CSP Orlando, Winter Park, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - University of Chicago Medical Center, Chicago, Illinois
  - Centennial Medical Group, Elkridge, Maryland
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - C.S. Mott Clinical Research Center (CRC), Detroit, Michigan
  - Beaumont Infectious Diseases Research, Royal Oak, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - CVS Health - Site 02815 East Brunswick, East Brunswick, New Jersey
  - Hackensack Meridian Jersey Shore University Medical Center, Neptune City, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Onsite Clinical Solutions (secondary location), Charlotte, North Carolina
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - WellNow Urgent Care and Research - Columbus, Columbus, Ohio
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Heritage Valley Multispecialty Group, Inc, Beaver, Pennsylvania
  - Premier Primary Care, Union City, Tennessee
  - Nayak Research, LLC, Andrews, Texas
  - Headlands Research - Brownsville, Brownsville, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Next Innovative Clinical Research, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - Accurate Clinical Research - East Humble, Humble, Texas
  - Accurate Clinical Research, Inc, Humble, Texas
  - Sun Research Institute, San Antonio, Texas
  - Eastside Research Associates, Redmond, Washington
- Canada (4):
  - Dawson Clinical Research, Guelph, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
  - Medical Trust Clinics, Oshawa, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario
- Greece (5):
  - Thoracic General Hospital of Athens "I Sotiria", Athens, Attica
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - Alexandra General Hospital of Athens, Athens, Attikí
  - General Hospital of Athens "Laiko", Athens
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
- Italy (4):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - ASST Fatebenefratelli Sacco, Milan, Milano
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Taiwan (4):
  - Far Eastern Memorial Hospital, New Taipei City, NEW Taipei
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Zhang W, Terra SG, Weinstein EA, Bramson C, Leister-Tebbe H, Baniecki ML, Guan S, Agyemang A, Antonucci S, Wisemandle W, Hammond J. Retreatment With Nirmatrelvir/Ritonavir Following Return of COVID-19 Symptoms and SARS-CoV-2 Positivity. Clin Infect Dis. 2025 Sep 30:ciaf548. doi: 10.1093/cid/ciaf548. Online ahead of print. PMID 41027009
- [Derived] Baniecki ML, Guan S, Rai DK, Yang Q, Lee JT, Hao L, Weinstein E, Hyde C, Cardin RD, Soares H, Hammond J. Integrated virologic analysis of resistance to nirmatrelvir/ritonavir in individuals across four phase 2/3 clinical studies for the treatment of COVID-19. EBioMedicine. 2025 Aug;118:105819. doi: 10.1016/j.ebiom.2025.105819. Epub 2025 Jun 30. PMID 40592258
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671042

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 436 participants were randomized and treated in this study with a repeat 5-day treatment course of nirmatrelvir/ritonavir or placebo/ritonavir for mild-to moderate coronavirus disease 2019 (COVID-19).
Groups:
- Nirmatrelvir 300 mg + Ritonavir 100 mg: Participants received nirmatrelvir 300 milligrams (mg) (participants with estimated glomerular filtration rate [eGFR] greater than or equal to [>=] 30 to less than [<] 60 milliliter per minute [mL/min]/1.73 meters squared [m^2] or estimated creatinine clearance [CrCl] >=30 to <60 mL/min received 150 mg every 12 hours [q12h] for 5 days) and ritonavir 100 mg, orally for 5 days q12h from Day 1 to Day 5.
- Placebo + Ritonavir 100 mg: Participants received placebo matched to nirmatrelvir followed by ritonavir 100 mg orally, for 5 days q12h from Day 1 to Day 5.
Period: Overall Study
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo + Ritonavir 100 mg
Started | 292 | 144
Completed | 280 | 138
Not Completed | 12 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants randomly assigned to study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo + Ritonavir 100 mg | Total
Number analyzed (Participants) | 292 | 144 | 436
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (16.52) | 53.5 (16.43) | 53.5 (16.47)
Age, Customized [Count of Participants; unit: Participants]
  12 to less than 18 years | 1 | 0 | 1
  18 to 44 years | 88 | 40 | 128
  45 to 64 years | 121 | 64 | 185
  >= 65 years | 82 | 40 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 80 | 247
  Male | 125 | 64 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 159 | 72 | 231
  Not Hispanic or Latino | 131 | 72 | 203
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 13 | 2 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 264 | 132 | 396
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 5 in Viral Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Ribonucleic Acid (RNA) Level in Nasopharyngeal (NP) Swabs: mITT Population
Description: Baseline was defined as the latest measurement between Day -1 and Day 1, but post-dose samples that were collected within 1 hour post start of dosing were also treated as baseline. Samples with result "< lower limit of quantification (LLOQ)" were imputed as 1.7 log10 copies/milliliter (mL), and samples with result "Not Detected" were imputed as 0.0 log10 copies/mL.
Time Frame: Baseline, Day 5
Population: Modified intent-to-treat (mITT) analysis population included all participants randomly assigned to study intervention who took at least 1 dose of study intervention and who had a positive viral RNA NP swab test result (>= 2.0 log10 copies per mL) at baseline. Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Log10 copies/mL
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo + Ritonavir 100 mg
Number analyzed (Participants) | 218 | 113
Log10 copies/mL | -3.871 (0.129) [lower limit 0.129] | -3.166 (0.171) [lower limit 0.171]
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo + Ritonavir 100 mg; Mixed model for repeated measures (MMRM) included fixed effects of treatment, geographic region, baseline SARS-CoV-2 RNA level, visit, and treatment-by-visit interaction; an unstructured (co) variance structure was used; Test type: Superiority; p = 0.0004, MMRM; Least square (LS) mean difference = -0.705, 95% CI 2-sided [-1.093 to -0.316]

2. Secondary Outcome: Time to Two Consecutive Negative Rapid Antigen Test (RAT) Results At Least 24 Hours Apart Through Day 28: mITT Population
Description: The event of 2 consecutive negative RAT results obtained at least 24 (-2) hours apart through Day 28 was defined as achieving 2 consecutive non-missing RATs with negative results through Day 28, where the 2 tests were at least 22 hours and at most 7 days apart. For the event of 2 consecutive negative RAT results obtained at least 24 hours apart through Day 28, the date of the first negative RAT result was considered the first event date. Time to 2 consecutive negative RAT results obtained at least 24 hours apart defined as: for participant achieving event, time to event = (first event date) -(first dose date) + 1. For participant not achieving event (censored), censoring date was at last date of RAT measurement, time = (censoring date) - (first dose date) + 1 or Day 27 whichever occurred first (Day 27 was last possible day to achieve 2 consecutive negative RAT results obtained at least 24 hours apart through Day 28).
Time Frame: Day 1 of dosing maximum up to Day 28 or censoring date, whichever occurred first
Population: mITT analysis population included all participants randomly assigned to study intervention who took at least 1 dose of study intervention and who had a positive viral RNA NP swab test result (>= 2.0 log10 copies per mL) at baseline. Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo + Ritonavir 100 mg
Number analyzed (Participants) | 223 | 115
Days | 4.000 [4.000 to 5.000] | 5.000 [5.000 to 6.000]
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo + Ritonavir 100 mg; Analysis was based on Cox proportional hazard (PH) model which included treatment, geographic region, baseline SARS-CoV-2 RNA level (< 4 log10 copies/mL or >= 4 log10 copies/mL) and time since the last vaccination (less than or equal to [<=6] months, > 6 months or unvaccinated) as appropriate; Test type: Superiority; p = 0.0697, COX proportional hazard ratio; Hazard Ratio (HR) = 1.235, 95% CI 2-sided [0.983 to 1.551]

3. Secondary Outcome: Time to Sustained Alleviation of All Targeted Signs and Symptoms Through Day 28: mITT Population
Description: Sustained alleviation of all targeted COVID-19 signs/symptoms was defined as the event occurring on the first of 2 consecutive days when all symptoms scored as moderate or severe at study entry are scored as mild or absent and all symptoms scored mild or absent at study entry are scored as absent. The first day of the 2 consecutive-day period was considered the first event date. The time to sustained symptom alleviation was defined as for a participant with sustained symptom alleviation, time to event was calculated as (First Event Date) - (First Dose Date) +1. For a participant that either completed Day 28 of the study or discontinued from the study before Day 28 without sustained symptom alleviation (censored), censoring date was at the last date on which symptom alleviation was assessed, and time was calculated as (Censoring Date) - (First Dose Date) +1 or Day 27 whichever occurred first.
Time Frame: Day 1 of dosing maximum up to Day 28 or censoring date, whichever occurred first
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo + Ritonavir 100 mg
Number analyzed (Participants) | 186 | 99
Days | 8.000 (7.000) [7.000 to 10.000] | 9.000 (8.000) [8.000 to 11.000]
Statistical Analysis 1: Comparison: Nirmatrelvir 300 mg + Ritonavir 100 mg vs Placebo + Ritonavir 100 mg; Analysis was based on Cox proportional hazard (PH) model which included treatment, geographic region, baseline SARS-CoV-2 RNA level (< 4 log10 copies/mL or >= 4 log10 copies/mL) and time since the last vaccination (<=6 months, > 6 months or unvaccinated) as appropriate; Test type: Superiority; p = 0.5202, COX proportional hazard ratio; Hazard Ratio (HR) = 1.084, 95% CI 2-sided [0.848 to 1.385]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Discontinuation From Study
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect, was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or nonpathogenic. TEAEs were defined as AE that started on or after study medication on Day 1 up to Week 24 follow-up. AEs included both SAEs and all non-SAEs.
Time Frame: Day 1 of dosing up to maximum Week 24 follow-up
Population: Safety population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo + Ritonavir 100 mg
Number analyzed (Participants) | 289 | 144
Participants
  AEs | 148 | 55
  SAEs | 3 | 1
  AEs leading to discontinuation from study | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to maximum Week 24 follow-up
Description: An event may be categorized as serious in 1 participant and non-serious in other, or a participant may experience both serious and non-serious event. Safety population: all participants randomly assigned to study intervention, who took at least 1 dose of study intervention.
Arm/Group | Nirmatrelvir 300 mg + Ritonavir 100 mg | Placebo + Ritonavir 100 mg
All-Cause Mortality (participants affected / at risk) | 0/289 | 0/144
Serious Adverse Events (participants affected / at risk) | 3/289 | 1/144
Other Adverse Events (participants affected / at risk) | 29/289 | 2/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirmatrelvir 300 mg + Ritonavir 100 mg (N=289) | Placebo + Ritonavir 100 mg (N=144)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirmatrelvir 300 mg + Ritonavir 100 mg (N=289) | Placebo + Ritonavir 100 mg (N=144)
Dysgeusia (Nervous system disorders) | 29 (29) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT05567952/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT05567952/SAP_001.pdf